CLINICAL TRIAL: NCT06851858
Title: A Phase II Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of AZD6234 in Participants Living With Overweight or Obesity With Type 2 Diabetes Who Are on a Stable Dose of GLP-1 Receptor Agonist
Brief Title: Efficacy, Safety and Tolerability of AZD6234 in Participants Living With Overweight or Obesity With Type 2 Diabetes Who Are on a Stable Dose of GLP-1 Receptor Agonist
Acronym: ARAY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D8750C00005
Record Dates: First submitted 2025-02-13; First posted 2025-02-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Endocrinology; Diabetes, Type II; Obesity
Keywords: Diabetes, Type II; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: The study spans approx. 37 weeks per participant, including a screening period, a treatment period and a follow-up period. Around 64 eligible participants will be randomized to receive either AZD6234 or a matching placebo, in addition to their stable GLP-1 RA regimen. Treatments consist of weekly subcutaneous injections, with AZD6234 dosing adjustments allowed based on individual tolerance.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study in which AstraZeneca, the study site staff, and participants remain blinded during the clinical study. All packaging and labelling of IMP will be done in such a way as to ensure blinding for all participants, AstraZeneca staff, and study site staff. Blinded investigators, blinded study site staff, and participants will remain blinded to each participant's assigned IMP throughout the course of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD6234 (Experimental): Weekly SC injections of AZD6234
  Interventions: Drug: AZD6234
- Placebo for AZD6234 (Placebo Comparator): Weekly SC injections of matching placebo
  Interventions: Drug: Placebo to match

INTERVENTIONS:
Drug: AZD6234 — Weekly SC injections of AZD6234
  Arms: AZD6234
Drug: Placebo to match — Weekly SC injections of matching placebo
  Arms: Placebo for AZD6234

SUMMARY:
This Phase II study is a randomized, parallel group, double blinded, placebo-controlled, multicenter to evaluate the efficacy, safety, and tolerability of AZD6234 in adults with overweight or obesity and type 2 diabetes on stable GLP-1 RA therapy.

DETAILED DESCRIPTION:
This is a Phase II, randomised, parallel-group, double-blind, placebo-controlled, multi-centre study to assess the efficacy, safety, and tolerability of AZD6234 compared with placebo, given once weekly as a subcutaneous (SC) injection, in adults living with overweight or obesity and type 2 diabetes who are on a stable dose of GLP-1 RA. The study is being conducted across sites in the USA to evaluate the efficacy, safety, and tolerability of AZD6234 in adults with overweight or obesity and type 2 diabetes on stable GLP-1 RA therapy. A total of 64 Participants, aged 18-75 with a BMI ≥ 27 kg/m², will be randomized to receive weekly subcutaneous injections of either AZD6234 or a placebo, alongside their current GLP-1 RA medication. The study involves a screening period and a treatment and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 75 years old at the time of signing the informed consent.
2. Diagnosed with type 2 diabetes ≥ 180 days before screening.
3. HbA1c value at screening of ≥ 6.0% (42 mmol/mol) and ≤ 10% (86 mmol/mol).
4. On a stable maintenance dose of an injectable GLP-1 RA.
5. At Screening, have a BMI ≥ 27 kg/m2

Exclusion Criteria:

1. Has received treatment with prescription or non-prescription medication for weight loss within the last 3 months prior to screening (other than a GLP-1 RA).
2. Self-reported weight change of > 5 % in the 3 months prior to screening.
3. Diabetes mellitus that is not clearly type 2 diabetes.
4. Use of insulin therapy for T2DM
5. Previous or planned (within study period) bariatric surgery or fitting of a weight loss device (eg, gastric balloon or duodenal barrier)
6. Significant hepatobiliary disease (except for non-alcoholic steatohepatitis or nonalcoholic fatty liver disease without portal hypertension or cirrhosis)

8. Impaired renal function defined as eGFR ≤ 45 mL/minute/1.73m2 at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight from baseline at Study Week 26 | From baseline to week 26
  To determine whether treatment with AZD6234 is superior to placebo for weight loss at Study Week 26
Weight loss ≥ 5% from baseline at Study Week 26 | From baseline to week 26
  To assess the effect of AZD6234 versus placebo on the proportion of participants with weight loss ≥ 5% from baseline at Study Week 26

SECONDARY OUTCOMES:
Weight loss ≥ 10% from baseline at Study Week 26 | From baseline to week 26
  To assess the effect of AZD6234 versus placebo on the proportion of participants with weight loss ≥ 10% from baseline at Study Week 26
Absolute change in body weight (kg) from baseline at Study Week 26 | From baseline to week 26
  To determine whether AZD6234 is superior to placebo for absolute weight reduction (kg) at Study Week 26
Change in HbA1c from baseline at Study Week 26. | From baseline to week 26
  To assess the effect of AZD6234 versus placebo on glycaemic control at Study week 26
AZD6234 plasma concentrations | From baseline to week 26
  To characterise the PK of AZD6234
Change in serum glucose from baseline at Study Week 26. | From baseline to week 26
  To assess the effect of AZD6234 versus placebo on glycaemic control at Study week 26

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Doral, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Canton, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Newton, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Kansas City, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Norman, Oklahoma
  - Research Site, Knoxville, Tennessee
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/